CLINICAL TRIAL: NCT05824195
Title: Evaluation of Potentially Bioactive Foods With Respect to Cardiometabolic- and Cognitive Test Variables
Brief Title: Evaluation of Potentially Bioactive Foods With Respect to Cardiometabolic Test Variables
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Anne Nilsson, Associate professor, Lund University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Dnr: 2019-00980
Record Dates: First submitted 2023-04-06; First posted 2023-04-21 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Healthy Subjects; Diet, Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Quinoa1 (Experimental): Quinoa bread type1.
  Interventions: Other: Bread products
- Quinoa 2 (Experimental): Quinoa bread type 2
  Interventions: Other: Bread products
- Quinoa 3 (Experimental): Quinoa bread type 3
  Interventions: Other: Bread products
- Reference (Sham Comparator): A white wheat bread
  Interventions: Other: Bread products

INTERVENTIONS:
Other: Bread products — Four intervention products were included in the study. Three experimental breads (quinoa 1, quinoa 2, quinoa 3) were developed, and consisted of white wheat breads substituted with the differrent quinoa types. The reference product included was a white wheat bread without quinoa. All intervention products contain 50 g available starch.

SUMMARY:
The overall goal is to increase the knowledge that can be used for the development of food products with antidiabetic properties, with the aim of facilitating healthier food choices for people. More specifically, the primary aim of this project is to evaluate the effects of different varieties of quinoa on postprandial glucose tolerance and subjective appetite markers. The crossover, randomised dietary intervention study will be conducted in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 20-28
* age between 18-40 years
* Healthy
* consume a diet in accordance with Nordic Nutrition Recommendations

Exclusion Criteria:

* not vegan
* metabolic diseases (such as diabetes)
* Gastro intestine tract problems or irritable bowel syndrome
* known food allergies of intolerances
* smoker
* antibiotics should not have been consumed during the last 4 weeks
* probiotics should not have been consumed during the last 4 weeks

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-06-03 (Actual); Study Completion 2023-06-03 (Actual)

PRIMARY OUTCOMES:
Glucose tolerance | 3 hours. Fasting (time =0 minutes), 15 minutes, 30 minutes, 45 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, 180 minutes
  Capillary blood glucose concentrations are measured repeatedly after test products consumed at breakfast. The postprandial incremental glucose area under the curve is used as a measure of glucose tolerance.

SECONDARY OUTCOMES:
serum insulin | 3 hours. Fasting (time =0 minutes), 15 minutes, 30 minutes, 45 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, 180 minutes
  Capillary serum insulin concentrations are measured repeatedly after test products consumed at breakfast. The postprandial incremental insulin area under the curve is used as a measure of insulin excretion needed for the control of the postprandial blood glucose increments.
Subjective appetite sensations (hunger, satiety, and desire to eat) | 3 hours. Fasting (time =0 minutes), 30 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, 180 minutes
  subjects will rank subjective appetite sensations repeatedly in the postprandial period after the test breakfasts, using 10 cm visual analogue scales.

CONTACTS AND LOCATIONS:
Locations (1):
- Lund University, dep of Food Technology, Engineering, and Nutrition, Lund, Välj..., Sweden

IPD SHARING:
Plan to Share IPD: No